CLINICAL TRIAL: NCT00170495
Title: Etiology and Impact of Acute Viral Respiratory Infections in Ambulatory Elderly Populations
Brief Title: Acute Viral Respiratory Infections in Elderly
Status: Terminated | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Robert Johnson, HHS/NIAID/DMID
Other Study IDs: 04-049; H-14802
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2008-09

CONDITIONS: Respiratory Infections, Acute
Keywords: respiratory illness, influenza, bronchitis, pneumonia, cold
MeSH Terms: conditions — Respiratory Tract Infections; Influenza, Human; Bronchitis; Pneumonia; Common Cold

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood, sputum, nasal and throat swabs

GROUPS / COHORTS (1):
- observation: male and female adults age 65 and older with acute respiratory illness (common colds, flu, bronchitis, pneumonia)

SUMMARY:
This study is designed to assess the causes and impact of acute respiratory illness (common colds, flu, bronchitis, pneumonia) in adults age 65 and older. One of the ways to determine the virus causing a particular illness is to get a blood specimen when a person is sick and again later and look for the body's specific responses that identify the virus. Approximately 3000 subjects will be evaluated and their medical records assessed for details of recent illness and general health to help in understanding the subjects' current illness.

DETAILED DESCRIPTION:
The purpose of this study is to determine the role of respiratory viruses in the etiology of medically attended acute respiratory illness in elderly populations and to assess the impact of these illnesses. Ambulatory elders presenting for health care with an acute respiratory illness will be recruited. Nose and throat swab specimens will be collected to test for one of the respiratory viruses, and acute and convalescent blood specimens will be collected to test for increases in specific antibody. Specimens will be collected within seven days of the onset of illness and then 1 month later for comparison specimens. A brief questionnaire will accompany the specimens, and more complete data on the illness and consequences will be obtained from the medical record. The pattern of illnesses by virus and their severity and duration will be determined.

ELIGIBILITY:
Inclusion Criteria:

1. 65 years of age or older
2. Presentation to the geriatric clinic with an acute respiratory illness of less than 7 days' duration.

Exclusion Criteria:

1. Presentation to the geriatric clinic with a history of a respiratory illness of greater than 7 days' duration.
2. Physician/physician assistant judgment that the respiratory complaints do not represent an acute infection.
3. Patient declines to permit specimen collection.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: male and female adults age 65 and older with acute respiratory illness (common colds, flu, bronchitis, pneumonia)
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2004-09; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States